CLINICAL TRIAL: NCT00572130
Title: A Phase II Study of Intravenous Rexin-G in Recurrent or Metastatic Osteosarcoma
Brief Title: Phase II Study of Intravenous Rexin-G in Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Epeius Biotechnologies (Industry)
Responsible Party: Erlinda M. Gordon, M.D., Epeius Biotechnologies Corporation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C07-110
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-02

CONDITIONS: Osteosarcoma
Keywords: Tumor-targeted gene medicine; Cyclin G1 gene; Osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rexin-G Dose 1 (Experimental)
  Interventions: Genetic: Rexin-G Dose 1
- Rexin-G Dose 2 (Experimental)
  Interventions: Genetic: Rexin-G Dose 2

INTERVENTIONS:
Genetic: Rexin-G Dose 1 — Rexin-G i.v., 1 x 10e11 cfu, two times a week x 4 weeks, rest 2 weeks May be repeated if grade 1 or less toxicity
  Arms: Rexin-G Dose 1
Genetic: Rexin-G Dose 2 — Rexin-G i.v., 1 x 10e11 cfu, three times a week x 4 weeks; rest 2 weeks May repeated if grade 1 or less toxicity
  Arms: Rexin-G Dose 2

SUMMARY:
Rexin-G is a tumor-targeted gene medicine that is designed to seek out and destroy both primary tumors and metastatic cancers without the side effects of standard chemotherapy. The objectives of the study are: (1) to evaluate the clinical effectiveness of intravenous injections of Rexin-G, a tumor-targeted gene vector, in controlling tumor growth and prolonging life, and (2) to evaluate its over-all safety.

DETAILED DESCRIPTION:
The adaptive trial design of this advanced Phase II study incorporates (i) a dosing schedule based on the patient's estimated tumor burden and not on standard dosing per kilogram body weight or body surface area, and (2) a tumor response evaluation process that is unique to the manner in which osteosarcoma responds favorably to therapy, i.e., with necrosis and increasing calcification in metastatic tumors and decreased glucose utilization using PET-CT imaging studies.

Twenty to thirty patients will receive Rexin-G at either Dose Level 1 or 2. Patients will be assigned a dose level based on the estimated tumor burden as measured by PET-CT imaging studies. Estimated tumor burden is measured by multiplying the sum of the longest diameters of target lesions in cm by 10e9 cancer cells. If the tumor burden is less than 10 billion cells, the patient will be assigned to Dose Level 1, if the tumor burden is greater than 10 billion cells, the patient will be assigned to Dose Level 2.

*Treatment Cycle Dose Level Vector Dose/Day Max.Volume/Dose

Two times a week 1 1.0 x 10e11 cfu 200 ml

Three times a week 2 1.0 x 10e11 cfu 200 ml

* Each treatment cycle will be six weeks (four weeks of treatment and two weeks of rest). Patients who have resolution of toxicity to < grade I may have repeat cycles. After one or more treatment cycles, the principal investigator may recommend surgical debulking or complete surgical removal. If residual disease is present either by histopathological examination or by PET-CT scan, repeat treatment cycles may be given 3-4 weeks after surgery, if the surgical incision has healed, and if the patient has < grade I toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with recurrent or metastatic osteosarcoma who is considered refractory to known therapies.
2. Histologically or cytologically confirmed osteosarcoma that is measurable.
3. Adequate hepatic function: Total bilirubin < 2.0 mg/dL (upper limit included); AST/ALT < 2x institutional norm; alkaline phosphatase < 2.5x upper limit of institutional norm unless the patient has extensive bone metastases. Patients with elevated alkaline phosphatase due to extensive liver disease will be excluded from study; albumin > 3.0 mg/dL. There must be no substantial ascites. PT and PTT must be within normal limits.
4. Performance status must be < 1 (ECOG 0-1) with a life expectancy of at least 3 months.
5. Hemoglobin > 9 gms%
6. Absolute granulocyte count > 1000/uL, and platelet count > 100,000/uL.
7. Serum creatinine of less than 1.5 mg%.
8. There must be no plans for the patient to receive further cancer therapy from the date of enrollment until the completion of the 6-week follow-up visit.
9. Accessibility of peripheral or central IV line
10. Age > 10 years
11. Patients will be off chemotherapy for a minimum of 4 weeks prior to initiation of therapy and should have recovered to Grade 1 or less toxicity.
12. The ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Prior malignancy, except for non-melanoma skin cancer, stage 1 breast cancer, CIS of cervix from which the patient has been disease-free for 5 years.
2. Woman who are pregnant or nursing
3. Fertile patients unless they agree to use barrier contraception (condoms and spermicide jelly) during the vector infusion period and for six weeks after infusion. Male patients must agree to use barrier contraception.
4. Patients who are transfusion dependent (more than one transfusion per month)
5. Patients with medical, psychiatric, or social conditions that would compromise successful adherence to this protocol.
6. Patient who do not meet the inclusion criteria.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-12; Primary Completion 2010-07 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy as measured by over-all response rates (either CR, PR or SD) by International PET criteria | 12-18 months

SECONDARY OUTCOMES:
Clinical efficacy as measured by progression-free survival greater than one month and over-all survival of 6 months or longer; clinical toxicity measures | 12-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Sant P Chawla, M.D., Principal Investigator — Epeius Clinical Research Unit/Sarcoma Oncology Center
Locations (1):
- Epeius Clinical Research Unit/Sarcoma Oncology Center, Los Angeles, California, United States

REFERENCES:
- See also: Sponsor's Official Website — http://www.epeiusbiotech.com